CLINICAL TRIAL: NCT01301664
Title: Cartilage Tissue Engineering
Status: Available | Type: Expanded Access
Sponsor: Chin-Hung Chang (Other)
Responsible Party: Sponsor-Investigator, Chin-Hung Chang, MD.PhD., Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Other Study IDs: 97022
Record Dates: First submitted 2010-10-05; First posted 2011-02-23 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Mesenchymal Stem Cells
Keywords: The bone marrow-derived mesenchymal stem cells (BMMSCs) were obtained from redundant bone marrow from drilling during the joint replacement surgery.; The synovial-derived mesenchymal stem cells (SMSCs) were isolated from synovial membranes in the joint replacement surgery.; Cartilage slices were obtained from discard cartilage in the joint replacement surgery.
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

INTERVENTIONS:
Other: total knee / hip replacement — Human cartilage tissues were harvested from osteoarthritic patient during total knee arthroplasty surgery.

SUMMARY:
In this study, the investigators explored the hypothesis that osteoarthritic cartilage fragments can promote chondrogenesis of MSCs. Non-wearing parts of cartilage tissues were harvested from one osteoarthritic patient during the total knee arthroplasty surgery. Cartilage fragments and MSCs were wrapped into fibrin glue; and the constructs were implanted subcutaneously into nude mice.

Moreover, the investigators will collect the discard cartilage to develop an acellular cartilage ECM-derived scaffold in the joint replacement surgery. In addition, the investigators will harvest the redundant bone marrow from drilling or useless synovium during the surgery to separate the mesenchymal stem cells. Furthermore, these mesenchymal stem cells will be transfected with hTERT for rejuvenation and then will be labeled with fluorescent dye PKH26 for application of animal study. To sum up, the investigators plan to use human, natural, and discard materials from the joint replacement surgery to develop appropriate allograft for cartilage repair and hope that one day this ideal would be apply in clinical.

DETAILED DESCRIPTION:
Extracellular matrix (ECM) is thought to participate significantly in guiding the differentiation process of mesenchymal stem cells (MSCs). In this study, we explored the hypothesis that osteoarthritic cartilage matrix can promote chondrogenesis of MSCs. Cartilage matrix was harvested from the health-like parts of osteoarthritic cartilage tissue. Cartilage fragments and MSCs were wrapped into fibrin glue; and the constructs were implanted subcutaneously into nude mice. Histological analysis showed a round and elongated cell appearance with positive Alcian blue staining of cartilage matrix formation in the constructs. However, the cells in fibrin glue only were condensed like MSCs in pellet culture. Immunohistochemical staining was abundantly positive for type II collagen in neo-cartilage regions of cartilage fragment-fibrin glue-MSC constructs, while the constructs without cartilage fragments were negative in staining for type II collagen. The gene expressions of type II collagen in the constructs with 60 mg fragments were significantly elevated after 4 weeks of implantation. Conversely, constructs without cartilage fragments failed to express type II collagen, which indicated that MSCs could not differentiate into a chondrogenic lineage. In conclusion, we demonstrated the effects of osteoarthritic cartilage matrix in promoting chondrogenic differentiation of MSCs. This was a favorable method without exogenous growth factors induction.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years old

Exclusion Criteria:

* more than 70 years old

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult